CLINICAL TRIAL: NCT00966433
Title: A Comparison of Different Ventilation Strategies in Children Using the Proseal™ Laryngeal Mask Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00009452
Record Dates: First submitted 2009-08-25; First posted 2009-08-27 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Intraoperative Ventilation
Keywords: Proseal™ LMA; children; ventilation; general anesthesia; Children under general anesthesia for outpatient surgery
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Spontaneous ventilation (Experimental): Pt's will be allowed to breathe spontaneously through the PLMA during surgery without the assistance of positive pressure ventilation.
  Interventions: Procedure: Spontaneous ventilation
- Pressure support ventilation (Experimental): Pt's will receive positive pressure assistance with each spontaneous breath through the PLMA.
  Interventions: Device: Pressure support Ventilation
- Pressure control ventilation (Active Comparator): Pt.'s will be placed on the ventilator and ventilated with pressure control. through the PLMA.
  Interventions: Device: Pressure control ventilation

INTERVENTIONS:
Procedure: Spontaneous ventilation — The patient will breathe spontaneously (on their own)while under general anesthesia throughout the duration of the surgery.
  Arms: Spontaneous ventilation
Device: Pressure support Ventilation — The patient will breathe on their own and with a little assistance from the anesthesia machine while under general anesthesia throughout the duration of the surgery.
  Arms: Pressure support ventilation
Device: Pressure control ventilation — The patient's ventilation will be completely supported by the anesthesia machine while under general anesthesia throughout the duration of the surgery.
  Arms: Pressure control ventilation

SUMMARY:
The purpose of this research study is to compare difference between breathing by oneself or with the partial help from an anesthesia machine in children under general anesthesia.

DETAILED DESCRIPTION:
The laryngeal mask airway (LMA) is a breathing device that sits above the vocal cords and allows the patient to breathe in and out adequately under general anesthesia (GA). The ProSeal™ LMA (PLMA™) is a specialized type of LMA with a design that permits the delivery of higher pressures to help the patient breathe in and out (ventilate) and also contains a channel to suction the stomach.

Children under GA may breathe through a PLMA in different ways. Spontaneous ventilation consists of the children breathing on their own through a PLMA™. Pressure support ventilation allows the patient to breathe on their own with additional help from the anesthesia machine. Pressure control ventilation allows the patient to breathe with the help of an anesthesia machine.

A child undergoing surgery requires a deep level of general anesthesia which negatively affects their ability to ventilate. Thus, children may not breathe in oxygen and carbon dioxide out adequately at this level of anesthesia and it may be beneficial to provide some level of support to enhance carbon dioxide exchange and to avoid hypoventilation.

This study will attempt to determine whether pressure support ventilation improves ventilation in children undergoing outpatient surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical classification 1,2 (Healthy or relatively healthy children)
* Subjects scheduled for outpatient surgical procedures.
* Surgical procedure anticipated to be < 90 minutes
* Subject weight of ≤ 20 kg (44 lbs)
* Subject age of 12 months to 5 years (inclusive)

Exclusion Criteria:

* Inpatient
* ASA physical classification of 3, 4 or E (sick children)
* Risk of aspiration
* Subjects with malignant hyperthermia or family history of malignant hyperthermia
* Subjects with tracheostomies

Ages: 12 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Templeton, M.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brain AI, McGhee TD, McAteer EJ, Thomas A, Abu-Saad MA, Bushman JA. The laryngeal mask airway. Development and preliminary trials of a new type of airway. Anaesthesia. 1985 Apr;40(4):356-61. PMID 4003736
- [Background] Mason DG, Bingham RM. The laryngeal mask airway in children. Anaesthesia. 1990 Sep;45(9):760-3. doi: 10.1111/j.1365-2044.1990.tb14449.x. PMID 2100990
- [Background] Shimbori H, Ono K, Miwa T, Morimura N, Noguchi M, Hiroki K. Comparison of the LMA-ProSeal and LMA-Classic in children. Br J Anaesth. 2004 Oct;93(4):528-31. doi: 10.1093/bja/aeh238. Epub 2004 Aug 6. PMID 15298876
- [Background] Lardner DR, Cox RG, Ewen A, Dickinson D. Comparison of laryngeal mask airway (LMA)- Proseal and the LMA-Classic in ventilated children receiving neuromuscular blockade. Can J Anaesth. 2008 Jan;55(1):29-35. doi: 10.1007/BF03017594. PMID 18166745
- [Background] Bagshaw O. The size 1.5 laryngeal mask airway (LMA) in paediatric anaesthetic practice. Paediatr Anaesth. 2002 Jun;12(5):420-3. doi: 10.1046/j.1460-9592.2002.00887.x. PMID 12060328
- [Background] Licina A, Chambers NA, Hullett B, Erb TO, von Ungern-Sternberg BS. Lower cuff pressures improve the seal of pediatric laryngeal mask airways. Paediatr Anaesth. 2008 Oct;18(10):952-6. doi: 10.1111/j.1460-9592.2008.02706.x. Epub 2008 Jul 21. PMID 18647269
- [Background] Wheeler M. ProSeal laryngeal mask airway in 120 pediatric surgical patients: a prospective evaluation of characteristics and performance. Paediatr Anaesth. 2006 Mar;16(3):297-301. doi: 10.1111/j.1460-9592.2005.01788.x. PMID 16490094
- [Background] Goldmann K, Jakob C. A randomized crossover comparison of the size 2 1/2 laryngeal mask airway ProSeal versus laryngeal mask airway-Classic in pediatric patients. Anesth Analg. 2005 Jun;100(6):1605-1610. doi: 10.1213/01.ANE.0000152640.25078.90. PMID 15920181
- [Background] Lopez-Gil M, Brimacombe J, Alvarez M. Safety and efficacy of the laryngeal mask airway. A prospective survey of 1400 children. Anaesthesia. 1996 Oct;51(10):969-72. doi: 10.1111/j.1365-2044.1996.tb14968.x. PMID 8984875
- [Background] Keidan I, Berkenstadt H, Segal E, Perel A. Pressure versus volume-controlled ventilation with a laryngeal mask airway in paediatric patients. Paediatr Anaesth. 2001 Nov;11(6):691-4. doi: 10.1046/j.1460-9592.2001.00746.x. PMID 11696145
- [Background] Lopez Gil ML, Brimacombe J, Clar B. Sevoflurane versus propofol for induction and maintenance of anaesthesia with the laryngeal mask airway in children. Paediatr Anaesth. 1999;9(6):485-90. doi: 10.1046/j.1460-9592.1999.00404.x. PMID 10597550
- [Background] Garcia-Fernandez J, Tusman G, Suarez-Sipmann F, Llorens J, Soro M, Belda JF. Programming pressure support ventilation in pediatric patients in ambulatory surgery with a laryngeal mask airway. Anesth Analg. 2007 Dec;105(6):1585-91, table of contents. doi: 10.1213/01.ane.0000287674.64086.f1. PMID 18042854

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Spontaneous Ventilation | Pressure Support Ventilation | Pressure Control Ventilation
Started | 11 | 11 | 11
Completed | 10 | 10 | 11
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spontaneous Ventilation | Pressure Support Ventilation | Pressure Control Ventilation | Total
Number analyzed (Participants) | 10 | 10 | 11 | 31
Age, Continuous [Mean (Standard Deviation); unit: Months] | 28 (18) | 32 (17) | 27 (16) | 28.9 (17.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3
  Male | 9 | 9 | 10 | 28
ASA Status [Count of Participants; unit: Participants] — A grade I is a normal healthy patient and a grade II is a patient with severe systemic disease
  Participants
    I | 9 | 8 | 9 | 26
    II | 1 | 2 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Differences in End-tidal Carbon Dioxide Compared Between the Spontaneous Ventilation and Pressure Support Ventilation Groups.
Description: Differences in End-tidal Carbon Dioxide Compared Between the Spontaneous Ventilation and Pressure Support Ventilation Groups will be calculated by subtracting the mean of End-tidal Carbon Dioxide from the PSV group to the SV group
Time Frame: up to 90 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Spontaneous Ventilation | Pressure Support Ventilation
Number analyzed (Participants) | 10 | 10
mmHg | 55.2 (5.5) | 47 (6)
Statistical Analysis 1: Comparison: Spontaneous Ventilation vs Pressure Support Ventilation; Test type: Other; p = .0051, t-test, 2 sided; Mean Difference (Final Values) = -8.2, 95% CI 2-sided [-13.61 to -2.79]

2. Primary Outcome: Differences Tidal Volume Compared Between the Spontaneous Ventilation and Pressure Support Ventilation Groups.
Description: Tidal Volume Compared Between the Spontaneous Ventilation and Pressure Support Ventilation Groups. Measured in mL/Kg and will be calculated by subtracting the mean of tidal volume from the PSV group to the SV group
Time Frame: up to 90 minutes
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Spontaneous Ventilation | Pressure Support Ventilation
Number analyzed (Participants) | 10 | 10
mL/kg | 4.0 (.8) | 7.6 (.5)
Statistical Analysis 1: Comparison: Spontaneous Ventilation vs Pressure Support Ventilation; Test type: Other; p = .0001, t-test, 2 sided; Mean Difference (Final Values) = 3.6, 95% CI 2-sided [2.97 to 4.23]

3. Primary Outcome: Mean Values of ETCO2 in SV and PCV Groups
Description: Mean Values of ETCO2 in SV and PCV groups reported in mmHg
Time Frame: up to 90 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Spontaneous Ventilation | Pressure Control Ventilation
Number analyzed (Participants) | 10 | 11
mmHg | 55.2 (5.5) | 43.1 (0.8)

4. Primary Outcome: Mean Tidal Volume Values Compared Between SV and PCV Groups
Description: Mean Tidal Volume Values compared between SV and PCV Groups. Measured in mL/kg
Time Frame: up to 90 minutes
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Spontaneous Ventilation | Pressure Control Ventilation
Number analyzed (Participants) | 10 | 11
mL/kg | 4.0 (0.8) | 7.6 (0.2)

5. Primary Outcome: Mean Values of ETCO2 Between the PSV and PCV Groups
Description: Mean Values of ETCO2 between the PSV and PCV Groups. Measured in mmHg
Time Frame: up to 90 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pressure Support Ventilation | Pressure Control Ventilation
Number analyzed (Participants) | 10 | 11
mmHg | 47.0 (6.0) | 43.1 (0.8)

6. Primary Outcome: Mean Values of Tidal Volume Between the PSV and PCV Groups
Description: Mean Values of Tidal Volume Between the PSV and PCV Groups. Measured in mL/kg
Time Frame: up to 90 minutes
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Pressure Support Ventilation | Pressure Control Ventilation
Number analyzed (Participants) | 10 | 11
mL/kg | 7.6 (0.5) | 7.6 (0.2)

7. Secondary Outcome: Differences in Respiratory Rates Between Spontaneous Ventilation and Pressure Support Ventilation Groups.
Description: Differences in respiratory rates between spontaneous ventilation and pressure support ventilation groups will be calculated by subtracting the mean of from the respiratory rates PSV group to the SV group.
Time Frame: up to 90 minutes
Measure: Mean (Standard Deviation); unit: breath/min
Arm/Group | Spontaneous Ventilation | Pressure Support Ventilation
Number analyzed (Participants) | 10 | 10
breath/min | 28.1 (5.3) | 14.2 (5.3)
Statistical Analysis 1: Comparison: Spontaneous Ventilation vs Pressure Support Ventilation; Test type: Other; p = .0001, t-test, 2 sided; Mean Difference (Final Values) = -13.9, 95% CI 2-sided [-18.88 to -8.92]

8. Secondary Outcome: Mean Values of Respiratory Rate Compared Between the Spontaneous Ventilation and Pressure Control Ventilation Groups.
Time Frame: up to 90 minutes
Measure: Mean (Standard Deviation); unit: breath/min
Arm/Group | Spontaneous Ventilation | Pressure Control Ventilation
Number analyzed (Participants) | 10 | 11
breath/min | 28.1 (5.3) | 21.2 (3.0)

9. Secondary Outcome: Mean Values of Respiratory Rate Compared Between Pressure Support Ventilation and Pressure Control Ventilation Groups.
Time Frame: up to 90 minutes
Measure: Mean (Standard Deviation); unit: breath/min
Arm/Group | Pressure Support Ventilation | Pressure Control Ventilation
Number analyzed (Participants) | 10 | 11
breath/min | 14.2 (5.3) | 21.2 (3.0)

ADVERSE EVENTS:
Time Frame: up to 90 minutes
Arm/Group | Spontaneous Ventilation | Pressure Support Ventilation | Pressure Control Ventilation
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No